# **HEROS Study**

## Human Epidemiology and Responses to SARS-CoV-2 Study

#### Information Sheet

# Hi HEROS families,

When you started the study the Information Sheet you read told you the study would last 24 weeks. We also asked you to collect 9 nose samples. More nose samples are collected if someone is sick. At that time, we didn't know that the COVID-19 virus would still be so active as we get close to the fall season. We are learning a lot from HEROS and would like to keep learning. We would like to see if there are any changes in how the COVID-19 virus spreads as we move into fall and winter. We are asking you and your family to continue in the study. We are asking each person to collect 4 more nose samples.

Just a reminder that at this time we are not able to give you any results from the tests that will be run. The samples that are collected will not be tested immediately; they will be stored and later run altogether. The laboratory that runs these tests is a research laboratory, and most research laboratories are not certified to report results for clinical purposes.

- Your participation is voluntary.
- You may ask questions at any time by contacting your study team.
- You may change your mind at any time.

# What you will need to do from your home.

In the beginning of the study we asked you to collect a nose sample every 2 weeks for 18 weeks (9 samples). We asked you to answer some questions on your phone, computer or over the phone each time you collect samples.

We are now asking if you and your family would collect 4 additional nose samples and answer questions just as you are doing now every 2 weeks.

# The last part of the study will now be at 28 weeks.

This visit may occur in your home or a visit to a medical center.

### **Payment**

Your family will continue to receive compensation based on how many samples you collect and study surveys you complete.

### A reminder that we are storing samples for future use.

The nose samples and blood samples that you collect will be used for genetic research to learn more about COVID-19. Your samples include your DNA. The DNA will only be used to study COVID-19. The genetic tests will study genes that are made up of DNA. Genes are present in each of the cells of your body and contain information needed for the human body to grow and function. Genes are passed down or "inherited" from parents to their children.

# **HEROS Study**

# Human Epidemiology and Responses to SARS-CoV-2 Study

### Information Sheet

**NOTE:** Your name will not be associated with the samples you provide. No one who works with the DNA will know that it is your DNA.

We understand that these are stressful times for you and your family. We thank you for your effort for the HEROS study. Please check yes below if you would like to continue in the extended study. If you check no, you will continue in the study and end at the regular date. If you would like more information, please check the option below and someone from your study site will contact you.

| Each member of your household who wishes to take part in this study has reviewed this information sheet and agrees to take part in the surveys and sample collections. |
|---|
| Yes, we want to continue in the study for a total of 28 weeks. We will collect the extra nose samples. |
| No, we do not want to do the extra 4 weeks. We want to complete the study for a total of 24 weeks |
| We would like more information before deciding |